CLINICAL TRIAL: NCT06521151
Title: The Effect of Audio Based Nutrition Education on Dietary Intake Practice, and Egg-based Diet Intervention on Nutrient Adequacy and Gestational Weight Gain Among Pregnant Women and Newborn's Birth Weights in the North Sidama Zone, Ethiopia.
Brief Title: The Effect of Audio Based Nutrition Education on Dietary Intake Practice, and Egg-based Diet Intervention on Nutrient Adequacy, and Gestational Weight Gain Among Pregnant Women and Newborn's Birth Weights in the North Sidama Zone, Ethiopia.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hawassa University (Other)
Collaborators: Ethiopian Public Health Institute (Other Government); Addis Ababa University (Other); Jima university (Unknown)
Responsible Party: Principal Investigator, Kaleb Mayisso Rodamo, Assistant professor, Hawassa University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB/098/16
Record Dates: First submitted 2024-06-02; First posted 2024-07-25 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Nutritional Deficiency
Keywords: Birth weight,
MeSH Terms: conditions — Malnutrition; Birth Weight

STUDY DESIGN:
Intervention Model Description: Following the baseline survey, four-arm cluster- randomized controlled trial (cRCT) will be conducted to evaluate the effectiveness of nutrition education and egg-based diet interventions on dietary intake practice, nutrient adequacy, and gestational weight gain among pregnant women and birth weight
Who Masked: Participant
Masking Description: A total of 300 pregnant women will be selected randomly from participants of the baseline survey, and enrolled in four arms in a 1:1:1:1 allocation ratios:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- egg based diet and Audio based nutrition education - group (arm-1) (Experimental): 76 pregnant women will be recruited to receive both egg based diet and audio based nutrition education
  Interventions: Dietary Supplement: egg based diet
- egg based diet alone- group (arm-2), (Experimental): 76 pregnant women will be recruited to receive egg based diet alone
  Interventions: Dietary Supplement: egg based diet
- Audio based nutrition education alone -group (arm- 3). (Experimental): 76 pregnant women will be recruited to receive audio based nutrition education alone
  Interventions: Dietary Supplement: egg based diet
- control arm (Arm-4) (No Intervention): 72 pregnant women will be employed in the control group to receive routine health education

INTERVENTIONS:
Dietary Supplement: egg based diet — egg based diet and audio based nutrition education group (arm-1), egg based diet alone group (arm-2), and audio based nutrition education alone group (arm- 3).
  Other Names: Audio based nutrition education
  Arms: Audio based nutrition education alone -group (arm- 3).; egg based diet alone- group (arm-2),; egg based diet and Audio based nutrition education - group (arm-1)

SUMMARY:
Background: Inadequate intake and utilization of nutrients during pregnancy is associated with inadequate nutrient adequacy and it has central implications on subsequent suboptimal weight gain and has an increased risk on low birth weight. Likewise, majority of Ethiopian pregnant women have inadequate nutrient intakes. These may be due to their poor dietary habits. Nutrition education is well-established intervention to enhance optimal dietary practices and is crucial to design appropriate diet interventions like multiple micronutrient and protein-energy supplements to optimize pregnancy outcomes.

However, in this country, integration of nutrition education with intervention of essential nutrients during pregnancy is not well studied. Therefore, this study is designed to measure the effect of nutrition education and egg-based diet interventions on dietary intake practice, nutrient adequacy, and gestational weight gain among pregnant women, and newborn's birth weight in North Sidama Zone.

Materials and methods: These studies will employee mixed study designs sequentially to address each specific objective. Baseline survey: A mixed method comprising community-based cross-sectional quantitative study complemented with a descriptive qualitative study that will be conducted in three woredas of North Sidama Zone in February 2024 to assess barriers and facilitators on the intake of adequate nutrients among pregnant women.

Following the baseline survey, four-arm cluster- randomized controlled trial (cRCT) will be conducted to evaluate the effectiveness of nutrition education and egg-based diet interventions on dietary intake practice, nutrient adequacy, and gestational weight gain among pregnant women and birth weight from March to August 2024. A total of 300 pregnant women will be selected randomly from participants of the baseline survey, and enrolled in four arms in a 1:1:1:1 allocation ratios: A multi-level mixed-effect logistic regression model will be used for quantitative data analysis, and a paired and independent t-test will be employed to measure the mean change in dietary intake practice, gestational weight gain and nutrient density between intervention and control groups. The qualitative data will be analyzed using Atlas-Ti software according to the inductive thematic content analysis approach.

Budget and work plan: For this study 1,102,200 ETB will be required. The study will be funded by Norad Project, Hawassa University, Sidama Regional Government and other possible grants in future. The study period will be March to August 2024.

ELIGIBILITY:
Inclusion Criteria:- .Pregnant women less and equal 12 weeks of pregnancy.

.Exclusion Criteria: Pregnant women who had been diagnosed with:-

* Confirmed hypertension
* Diabetes mellitus

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2024-05-31 (Actual); Primary Completion 2024-09-10 (Actual); Study Completion 2024-10-10 (Actual)

PRIMARY OUTCOMES:
Dietary Intake Practice | through study completion, an average of 1 month
  Dietary intake practice of pregnant women will be measured through assessing traditional and cultural beliefs (dietary intake habits, rituals, beliefs, values), pregnant woman's lifestyle (physical activity (type/frequency), alcohol intake and smoking practice, frequency of dining out, previous diet education, interest in dietary change, medicine use, usual and current appetite, weight history and meal pattern will be measured after delivery of audio based and banner prepared nutrition messages two times a month starting from second until the end of third trimester of pregnancy amongst pregnant women using standardized questionnaires•

SECONDARY OUTCOMES:
Gestational weight gain | through study completion, an average of 1 month,
  Gestational weight will be assessed through measuring the weight of the women using platform beam balance scale with movable weights or on a high-quality electronic scale. The scale should be graduated to the nearest 100 g (0.25 lb) and calibrated periodically against a known weight or series of weights approximating the range of weights encountered in clinic patients. The fewer clothes the better, as long as the weight of the clothing can be kept relatively constant for all women and all seasons of the year. This requires weighing women without purses, shoes, boots, coats, jackets, or any accompanying young children. All personnel responsible for taking weights and other measurements will be trained in the standard procedures. Optimal weight gain will be classified as: Normal weight women gain 17-25 kg at term, overweight women should gain 14-23 kg at term and obese women should gain 11-19 kg at term.
Adequacy of serum folate and iron | through study completion, an average of 1 week,
  serum level of folate and iron will be measured after dietary intervention of egg based diet during second and third trimesters of the pregnancy

OTHER OUTCOMES:
birth weight of new borne babies | through study completion, an average of 1 month,
  Birth weight will be assessed through accurate measurement of newborns to be weighed within an hour of birth using a well-calibrated scale measuring in 10 g increments. To prevent cross-infection, a thin clean cloth or paper will be placed on the scale. The device will be zeroed, the newborn will be placed on the scale naked, and the weight will be allowed to stabilize before being captured and recorded. We will classify the birth weight as 2500 grams extremely low birthweight: less than 1,000 grams (up to and including 999 grams), very low birthweight: less than 1,500 grams (up to and including 1,499 grams), low birthweight: less than 2,500 grams (up to and including 2,499 grams) and normal (birth weight ≥2.5 kg < 4.0 kg), or too heavy (macrosomia) (birth weight ≥ 4.0 kg)

CONTACTS AND LOCATIONS:
Locations (1):
- Hawassa University, Awasa, Sidama Region, Ethiopia

IPD SHARING:
Plan to Share IPD: Yes
all will be available up on resealable requested
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: September /2025

REFERENCES:
- [Derived] Mayisso K, Bosha T, Tamiru D. Effect of nutrition intervention coupled with healthy dietary advice on the nutritional status of pregnant women in the northern zone of the Sidama region, Ethiopia: a multilevel, cluster randomized controlled trial. J Health Popul Nutr. 2025 Jul 3;44(1):230. doi: 10.1186/s41043-025-00968-2. PMID 40611339
- See also: my closest colligue — http://amanuelyoseph45@gmail.com